CLINICAL TRIAL: NCT01837173
Title: Can Extracapsular Lymph Node Involvement be a Tool to Fine-tune UICC TNM 7th Edition for Esophageal Carcinoma?
Brief Title: Multicentric Retrospective Review of Extracapsular Lymph Node Involvement After Esophagectomy
Acronym: ECLNI-MC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, RN, MSc, Datamanager, University Hospital, Gasthuisberg
Other Study IDs: ECLNI-MC2013
Record Dates: First submitted 2013-04-02; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Cancer
Keywords: Adenocarcinoma; Squamous Cell Carcinoma; Neoadjuvant treatment; Esophagectomy
MeSH Terms: conditions — Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extracapsular LNI: Patients with positive lymph nodes that show extracapsular lymph node involvement
- Intracapsular LNI: Patients with positive lymph nodes that show NO extracapsular lymph node involvement

SUMMARY:
It is well known that lymph node metastasis is one of the most important prognostic factors in oesophageal carcinoma.

The investigators want to determine the influence of lymph node characteristics, being either intracapsular or extracapsular, on overall survival after esophagectomy for esophageal cancer.

DETAILED DESCRIPTION:
The classification of carcinoma of the esophagus has undergone a major modification between the UICC sixth (TNM-6) and TNM-7 edition. Regional lymph nodes (N) are now subdivided by the number of involved lymph nodes (pN0, 0; pN1, 1-2; pN2, 3-6; pN3 > 6), and distant metastasis (M) has been simplified to M1 rather than subdivided by location [1].

Nevertheless, TNM-7 doesn't take into consideration the morphologic characteristics of the metastatic lymph node itself. Since our first publications showing a negative relationship between presence of extracapsular lymph node involvement (EC-LNI) and survival [2], little has been published about the prognostic impact of this specific characteristic .

In our latest publication "Can extracapsular lymph node involvement be a tool to fine-tune pN1 for adenocarcinoma in UICC TNM 7th Edition?" [3], the investigators found a significant survival benefit for adenocarcinoma without extracapsular lymph node involvement in pN1 (= 1-2 positive lymph nodes) as compared to N2-N3 disease, treated by primary surgery. Moreover, pN1 patients with extracapsular lymph node involvement (EC-LNI) showed a survival that was comparable to patients with more than 2 positive lymph nodes (i.e. stage IIIB). These findings may have important consequences for future TNM adaptations.

The aim of this study is to validate our results on a larger, multicentric cohort, and if possible make recommendations and possible fine-tuning for a future TNM adaptation, including the characteristics of the metastatic lymph node itself, being intra- or extracapsular.

Furthermore the investigators want to examine if these effects are valid in pre-treated patients, i.e. surgery after neoadjuvant chemo(radiation) therapy. Although these patients are not incorporated in the current TNM classification, future adaptations to the TNM classification system will also examine the effects of neoadjuvant therapy (cfr. Rice/Blackstone WECC -Worldwide Esophageal Cancer Collaboration).

ELIGIBILITY:
Inclusion Criteria:

* Adequate lymph node sampling is of paramount importance. (pT1 - min. 10 LN; >pT2 min. 20 LN resected). At least the following lymph node stations should be examined: perioesophageal distal 1/3 and perigastric LN, left gastric artery, splenic artery, common hepatic artery, subcarinal lymph nodes. Sugical technique (transthoracic, transhiatal or minimal invasive) is less important if the criterium of adequate lymph node sampling is fulfilled but should be mentioned.

Exclusion Criteria:

* unforeseen organ metastasis
* subcardia tumors
* histology other than adenocarcinoma or squamous cell carcinoma
* Postoperative (inhospital or 30-day) mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric cohort study, patient chart analysis Since several high volume European institutions have published their results on patients with extracapsular lymph node involvement, we plan a pooling of their 'raw' data regarding type of treatment, histology, extracapsular LNI and (disease-free) survival.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival by LN-status (being ECLNI or ICLNI) | 5 yrs from surgery
  according UICC TNM7 pN (pN1-2-3)
Cancer-specific survival by LN-status (being ECLNI or ICLNI) | 5 yrs from surgery
  according UICC TNM7 pN (pN1-2-3)- censoring non-esophageal cancer related deaths

SECONDARY OUTCOMES:
Cancer specific survival for intra- and extracapsular lymph node involvement | 5 yrs from surgery
  Differentiation of intra- and extracapsular lymph node involvement after neoadjuvant chemo(radio)therapy followed by surgery versus primary surgery

OTHER OUTCOMES:
Cancer specific survival for intra- and extracapsular lymph node involvement | 5 yrs from surgery
  Differentiation of intra- and extracapsular lymph node involvement by histology, being Adenocarcinoma or Squamous cell carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Gasthuisberg, Leuven, Belgium